CLINICAL TRIAL: NCT01946750
Title: Predictive Value of the Immune Response of the Host in Clostridium Difficile Infections
Acronym: SERODIFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Versailles Hospital (Other)
Collaborators: Institut Pasteur (Industry); Sanofi Pasteur, a Sanofi Company (Industry); Saint Antoine University Hospital (Other)
Responsible Party: Principal Investigator, Alban LE MONNIER, Microbiological coordinator, Versailles Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P11/51_SERODIFF
Record Dates: First submitted 2012-12-20; First posted 2013-09-20 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections | interventions — Defecation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Case (Experimental): Hospitalized patient with clinical signs of Clostridium Difficile Infection and specific detection in stools of Clostridium Difficile toxins
  Interventions: Biological: Serum; Biological: Stools; Biological: Saliva; Biological: Whole blood
- Non-diarrheal control (Other): Hospitalized patient and asymptomatic carrier of Clostridium Difficile
  Interventions: Biological: Serum; Biological: Stools; Biological: Saliva; Biological: Whole blood

INTERVENTIONS:
Biological: Serum
Biological: Stools
Biological: Saliva — Optional sample collected for the cases and non-diarrheal control at the same time as the serum, to compare the presence of specific salivary Immune globulin type A (IgA) of C. difficile antibodies than in the serum.
Biological: Whole blood — Optional sample collected for the cases and non-diarrheal control at the same time as the serum, in order to study cellular immunity and describe the determinants of the development of a protective adaptive response.

SUMMARY:
Hypothesis: the antibody directed against certain antigens of Clostridium difficile would be predict the Clostridium difficile infection.

This study evaluates the weight of immunity by studying patients with Clostridium difficile infection versus controls (each patient is associated with two controls : diarrheal control without Clostridium difficile, and non-diarrheal control with or without Clostridium difficile). Recurrence and the kinetics of immune response following infection Clostridium difficile are studied by following the patients during three months.

There are also building biological samples collections clinically documented: sera, stool and strains.

ELIGIBILITY:
CASES :

Inclusion criteria of the cases :

* Hospitalized patients with clinical signs of Clostridium Difficile Infection and specific detection in stools of Clostridium Difficile toxins or/and isolating in stools and by digestive biopsy a strain producer of Clostridium Difficile toxins.
* Patients for which a serum prior to the episode of Clostridium Difficile Infection, ideally as far as possible of the episode, but at least 6 days before the day of diagnosis (D0) will be available.
* Patients for which consent has been signed or by their legal representative by default.
* Patients for whom is found Clostridium Difficile Infection in their file surgical and those for whom Clostridium Difficile Infection is the reason for admission will be included in the study but will be subject of a separate analysis, and their witnesses.

Exclusion criteria of the cases :

* Eligible patients for whom Clostridium Difficile Infection has been strongly suspected clinically but for which no microbiological confirmation will have been obtained.
* Eligible patients for whom no previous serum will have been recovered according to the criteria and conditions. The availability of a serum corresponding to the patient's admission is optional and can not be an exclusion criteria.
* Eligible patients (or their legal representatives) who are opposed to the use of their samples, the achieving samples and/or the longitudinal follow-up.
* Eligible patients who underwent plasmapheresis or treated with monoclonal antibodies to toxin A and B or immunoglobulins during the year preceding the episode of Clostridium Difficile Infection.
* Eligible patients but already included in the study for a recent infection with Clostridium Difficile or transferred to a second health facility for the same episode of Clostridium Difficile Infection.
* Eligible patients whose physicians responsible for the management refused participation in the study.
* Protected persons: pregnant women and children under the age of 18.

Secondarily be excluded the following cases:

* Patients for whom no sample has been achieved or retained by the laboratory of Medical Biology who participated in the diagnosis and monitoring of the patient.
* Hospitalized patients at the time of Clostridium Difficile Infection suspicion and diagnostic sample but released or transferred before rendering necessary microbiological results at baseline (J0 or J3).
* Matched control in a case excluded will be excluded.

NON-DIARRHEAL CONTROL : Eligible patients are those who do not have diarrhea at the time of recruitment.

To ensure that exposure to risks similar for cases and controls (hospitalization, usually care epidemic period, ...) will be recruited eligible patients according to the following criteria:

* Within a maximum period of six months after the inclusion of cases.
* Hospitalized in the same hospitalization service type as the case.
* With a duration of prior hospitalization at least as long as the time between admission and the corresponding case J0,
* Matched on sex and three age categories (18-40, 41-60 and> 60 years).

The inclusion of these controls depends on the one hand signing an informed consent for participation in the study and secondly the lack clinical signs suggestive of Clostridium Difficile Infection at the time of inclusion and known history of Clostridium Difficile Infection in their medical records (one no-diarrheal control hospitalized (ND) for one case).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Serum antibody titers | J-6, J0
  Consider the differential distribution of serum antibody titers, comparing experimental cases's sera prior episodes of Clostridium difficile infection (J-6) and the hospitalized controls's sera (J0).

SECONDARY OUTCOMES:
Kinetics of antibody | J-6, J0, J21, J90 and each recurrence
  The sera will be included in the analysis of the kinetics appearance of the immune response.
Clinical evolution | J90
  Cases and controls : patients will be followed for 3 months to monitor the clinical evolution (or death) after the of Clostridium difficile infection episode and determine the occurrence of any recurrence up to 3 months after the diagnosis.
Antibody titers for each antigen selected | J0
  Comparison of antibody titers for each antigen will be selected among different population groups formed : patients with Clostridium difficile infection, asymptomatic carriers patients, non-carriers patients including non-diarrheal and diarrheal (diarrhea due to other causes than Clostridium difficile infection).
Risk factors | 3 months
  Matching of controls on sex, type of service, age and length of hospital stay.
Molecular typing of Clostridium difficile strains | J0 and each recurrence
  Molecular characterization of strains isolated from patients with Clostridium difficile infection (experimental cases) and recurrence, to confirm microbiologically the notion of recurrence after a previous episode or occurrence of a new episode following infection by a new strain of Clostridium difficile.

CONTACTS AND LOCATIONS:
Overall Officials: Alban LE MONNIER, Microbiological coordinator, Principal Investigator — Versailles Hospital; Alix GREDER-BELAN, Clinical coordinator, Principal Investigator — Versailles Hospital
Locations (24):
- France (24):
  - CH Annecy Genevois, Annecy
  - Hôpital Jean Verdier, Bondy
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Hôpital Côte de Nacre, Caen
  - Hôpital Antoine Béclère, Clamart
  - CHU de Dijon - Hôpital d'Enfants, Dijon
  - Hôpital Raymond Poincaré, Garches
  - CHU de Grenoble, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - CHRU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - Hôpital Central de Nancy, Nancy
  - Fondation Hospitalière Sainte-Marie, Paris
  - Groupe Hospitalier Paris Saint Joseph, Paris
  - Groupe Hospitalier Sainte-Périne / Rossini / Chardon Lagache, Paris
  - Hôpital Lariboisière, Paris
  - Hôpital Saint Antoine, Paris
  - CHU de Reims - Hôpital Robert Debré, Reims
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen
  - CHU de Toulouse - Hôpital Purpan, Toulouse
  - CH de Tourcoing - Hôpital Gustave Dron, Tourcoing
  - CHRU de Tours - Hôpital Bretonneau, Tours
  - CH de Valenciennes, Valenciennes
  - Centre Hospitalier de Versailles, Versailles

IPD SHARING:
Plan to Share IPD: No